CLINICAL TRIAL: NCT03681821
Title: Effects of Transtheoretical Model-based Intervention on the Self-management of Patients With an Ostomy: a Randomized Controlled Trial
Brief Title: Effects of Transtheoretical Model-based Intervention on the Self-management of Patients With an Ostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Shali Wen, Principal investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: JLI
Record Dates: First submitted 2018-09-14; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Self-management; Self Efficacy
Keywords: ostomy; self-management; self-efficacy; health-promoting behavior
MeSH Terms: conditions — Health Behavior | interventions — Transtheoretical Model

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group had access to conventional care, in addition to receiving the follow-up TTM-based intervention sessions. The intervention was provided by trained nurses, including one researcher and one ET nurse. The researcher was regarded as primary leader of the intervention sessions. The leader informed patients of the schedule for each session using the educational manual 'we all can do the same: a pro-change program for self-management of an ostomy' (developed by psychologists, nursing managers, experienced ET nurses, and researchers).
  No interventions were performed for the control group participants during the study. However, these patients received conventional care in the colorectal surgery units according to the three hospitals' similar nursing guidelines.
Who Masked: Participant, Outcomes Assessor
Masking Description: Potential eligible participants were identified by researchers according to medical records at the colorectal surgery unit in each hospital. They were recruited with informed consent, and researchers explained the study purposes, procedures, benefits, and risks involved orally. The participants were then randomly allocated to the intervention or the control group according to a computer-generated block randomization list. The generated random numbers were put into consecutively numbered and opaque sealed envelopes. When enrolling and randomising a new participant, the enrolling investigators opened the sealed envelope after participant's name was written on next available envelopes. A sequentially numbered and opaque , sealed envelope system was used by a non-investigator. Additionally, all data collection was conducted by another research assistant who was blind to the study design and allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): Patients in the intervention group receiving the follow-up TTM-based intervention sessions.
  Interventions: Behavioral: Transtheoretical Model (TTM)-based Intervention
- The control group (No Intervention): No interventions except conventional care were performed for the control group.

INTERVENTIONS:
Behavioral: Transtheoretical Model (TTM)-based Intervention — Patients in the intervention group had access to conventional care, in addition to receiving the follow-up TTM-based intervention sessions. The intervention was provided by trained nurses, including one researcher and one ET nurse. Sessions were held in the meeting room in the unit four times: at baseline (T0), 2 days before discharge (T1), and at 1-month (T2) and 3-months (T3) after discharge, according to the assessment of their current stage of change delivered by filling the Stages of Change Subscale. Each face-to-face group contact lasted about 1 hour, depending on the complexity of the patients' problems.
  Arms: The intervention group

SUMMARY:
Colorectal cancer (CRC) is one of the most commonly diagnosed cancers worldwide. The main treatment approach is radical surgery, and the auxiliary treatment may be chemotherapy, radiotherapy, immunotherapy and other supportive therapies, which can increase the resection rate, reduce the recurrence rate, and improve the survival rate. Abdominoperineal resection with an ostomy and the formation of a permanent ostomy continue to be the primary and radical surgical approaches for many patients with rectal cancer, which results in the loss of defecation control function.

Although ostomy-related surgery is a life-saving procedure in most cases, it inevitably elicits some complex and lifelong consequences, such as uncontrolled gas and stool emissions, disturbed patients' body images, and effects their social and sexual lives, which place heavy pressure on ostomy self-management.

Some studies have revealed the various ways that patients' lives are affected by their stoma, including changes to their quality of life, body image, and social life, requiring coping and practical adjustments. Others have shown that not enough attention has been paid to patients' self-management abilities, with most care being provided by nurses or caregivers, leaving little opportunities for patients to manage on their own. Consequently, their self-management ability after discharge remains weak, especially their related knowledge and skills. Studies have shown that 33.0-80.4% of patients with an ostomy cannot cope with the problems encountered in ostomy care.

Many scholars focused on the ability of early self-management in patients with an ostomy after discharge, and there were several issues in the field of stoma nursing care, such as insufficient discharge preparedness because of shortened hospital stays and a lack of systematic acquisition of related knowledge and skills. Others highlighted the paucity of attention paid to the post-discharge needs of patients with a stoma and a lack of formal training for follow-up.

Currently, self-management programs for patients with an ostomy mainly focus on the passive problem-solving model led by nurses and less emphasize has been placed on the self-assessment of patients who passively accept relevant knowledge and skills. This is insufficient for the pertinence, continuity, operability, and promotion of self-management. It is essential to call for a patient-tailored and theoretical approach to improve self-management and promote rehabilitation.

The transtheoretical model (TTM) is an empirically validated model of individual behavioral change, which involves progress through a series of stages to make a particular behavioral change. TTM-based interventions have been applied to facilitate health behavioral changes, such as physical exercise, smoking cessation, and weight management, studies of which continue to demonstrate positive effects. There have been few studies of patients with an ostomy using TTM as an interventional tool to provide continuous and dynamic education. Therefore, this study decided to investigate the use of an integrated method of incorporating TTM into patient instruction and to provide assistance to enhance the self-management ability of patients with an ostomy.

The aim of this study was to determine the effects of a transtheoretical model (TTM)-based intervention on ostomy self-management on patients' stages of change, processes of change, decisional balance, and self-efficacy. The study's hypotheses were: (1) There would be no significant difference between the intervention group and the control group before the intervention, and after intervention there would be more patients in the intervention group than those in the control groups. (2) Patients in the intervention group would achieve greater improvement in the ability of self-management than those in the control group.

This study was a randomized controlled trial according to the CONSORT guidelines. The sample comprised 55 men and 37 women (24 to 77 years old, mean ± standard deviation = 52.8 ± 11.13 years). The study settings included three tertiary hospitals in Changsha, Hunan, China. The 92 patients recruited were randomized into a control group and an intervention group. Instruments, including self-management behaviors, were assessed at the baseline, 2 days before discharge and after 1-, 3- and 6-month follow-up. The chi-squared test, independent sample t test, and repeated-measures analysis of variance were used to analyze the data.

DETAILED DESCRIPTION:
The study was a single blind, follow-up, randomized, controlled trial. Researchers recruited subjects from three Central South University-affiliated general tertiary hospitals in Changsha, Hunan province, China. And the whole trail was on the basis of the CONSORT statements. These three hospitals provided similar conventional care for patients with an ostomy. Study procedures were approved by the institutional review boards of all participating centers before data collection began. All patients were screened by researchers for eligibility and then enrolled in the study if eligible and if the provided consent.

Potential eligible participants were identified by researchers according to medical records at the colorectal surgery unit in each hospital. They were recruited with informed consent, and researchers explained the study purposes, procedures, benefits, and risks involved orally. The participants were then randomly allocated to the intervention or the control group according to a computer-generated block randomization list. A sequentially numbered and opaque , sealed envelope system was used by a non-investigator.

The generated random numbers were put into consecutively numbered and opaque sealed envelopes. When enrolling and randomising a new participant, the enrolling investigators opened the sealed envelope after participant's name was written on next available envelopes; the enrolling investigators were blinded to the trial design and study hypotheses.

Patients in the intervention group had access to conventional care, in addition to receiving the follow-up TTM-based intervention sessions. The intervention was provided by trained nurses, including one researcher and one enterostomal therapy (ET) nurse. The researcher was regarded as primary leader of the intervention sessions. The leader informed patients of the schedule for each session using the educational manual'All can do the same: a pro-change program for self-management of an ostomy' (developed by psychologists, nursing managers, experienced ET nurses, and researchers).

Sessions were held in the meeting room in the unit four times: at baseline (T0), 2 days before discharge (T1), and at 1-month (T2) and 3-months (T3) after discharge, according to the assessment of their current stage of change delivered by filling the Stages of Change Subscale.

No interventions were performed for the control group participants during the study. However, these patients received conventional care in the colorectal surgery units according to the three hospitals' similar nursing guidelines. Preoperative visits for brief psychological counseling and general postoperative health education for ostomy cleaning, stoma appliance use, and self-care skills were provided by ward nurses. Additionally, post-discharge telephone follow-up focused on an unstructured interview and general health inquiries. To minimize contamination bias, the health education was implemented to avoid simultaneous scheduling for the two groups.

Data were collected by a research assistant who was blind to the study design and allocation of participants. At baseline, before randomization, socio-demographic and clinical characteristics were collected from medical records and personal interviews. The two groups of participants completed surveys after each follow-up via face to face interviews at baseline (T0), 2 days before discharge (T1), and at 1-month (T2) and 3-months (T3) after discharge. The last evaluation of scales was performed at 6-months (T4) of follow-up via telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Had received surgical treatment with a permanent ostomy for the first time;
* Must be Conscious, with normal communication ability;
* Must be volunteered to join the study.

Exclusion Criteria:

* Share a hospital room with a current study participant;
* With other types of cancer;
* Alcoholics and/or drug addicts;
* Disabilities and cannot take care of themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2013-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline the stages of change at 3 months | 3-months (T3) after discharge
  There were four subscales in the study, the stages of change subscale, the processes of change subscale, the decisional balance subscale, and the self-efficacy subscale.
  The outcome 1 was measured by the stages of change subscale and aimed to determine changes from baseline the percentage of participants of stages of change at 3 months. This subscale consisted of one item: 'Would you participant in self-management behavior of ostomy regularly?), which assess the patients' stages of self-management behavioral change, with five statements representing each stage: precontemplation, contemplation, preparation, action, and maintenance. Patients were asked to select one suitable statement that exactly described their current condition of ostomy self-management .
Change from baseline the scores of the processes of change at 3 months | 3-months (T3) after discharge
  The outcome 2 was measured by the stages of change subscale and aimed to determine changes from baseline the scores of the processes of change subscale at 3 months. This subscale was used to assess whether patients have had any activities or experiences that can affect their self-management of ostomy. It comprised 23 items and two dimensions, including cognitive level and behavioral level. Each individual item was scored from 1 (never) to 5 (always), with higher scores indicating higher frequency use of the process. The Cronbach values of the two dimensions were 0.958 and 0.905 respectively.
Change from baseline the scores of decisional balance at 3 months | 3-months (T3) after discharge
  The outcome 3 was measured by the stages of change subscale and aimed to determine changes from baseline the scores of decisional balance subscale at 3 months. This subscale was developed to assess patients' various points of view on the method of ostomy self-management that they had undertaken. It covered two dimensions of 20 items including perceived benefits and perceived barriers. Each item was ranked on a five-point Likert scale ranging from 1 (absolutely disagree) to 5 (absolutely agree). A higher score indicates a greater degree of agreement. The Cronbach's value of the perceived benefits and perceived barriers were 0.895 and 0.717, respectively.
Change from baseline the scores of self-efficacy at 3 months | 3-months (T3) after discharge
  The outcome 4 was measured by the stages of change subscale and aimed to determine changes from baseline the scores of self-efficacy subscale at 3 months. The scale consisted of eight items and aimed to assess patients' confidence in self-management. Each item is evaluated on a Likert-type scale (1-5). A higher score indicated stronger self-confidence. In this study, the Cronbach's coefficient level of the scale was 0.966 .

IPD SHARING:
Plan to Share IPD: No
The process of data collection cost a lot of human and material resources, some of the data was privacy information of participants, and so on. Considering this, it is improper to share these data.

REFERENCES:
- [Background] Ang SG, Chen HC, Siah RJ, He HG, Klainin-Yobas P. Stressors relating to patient psychological health following stoma surgery: an integrated literature review. Oncol Nurs Forum. 2013 Nov;40(6):587-94. doi: 10.1188/13.ONF.587-594. PMID 24161637
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421
- [Background] van Leer E, Hapner ER, Connor NP. Transtheoretical model of health behavior change applied to voice therapy. J Voice. 2008 Nov;22(6):688-98. doi: 10.1016/j.jvoice.2007.01.011. Epub 2007 Dec 21. PMID 18082367
- [Background] McGuire S. World Cancer Report 2014. Geneva, Switzerland: World Health Organization, International Agency for Research on Cancer, WHO Press, 2015. Adv Nutr. 2016 Mar 15;7(2):418-9. doi: 10.3945/an.116.012211. Print 2016 Mar. No abstract available. PMID 26980827
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Popek S, Grant M, Gemmill R, Wendel CS, Mohler MJ, Rawl SM, Baldwin CM, Ko CY, Schmidt CM, Krouse RS. Overcoming challenges: life with an ostomy. Am J Surg. 2010 Nov;200(5):640-5. doi: 10.1016/j.amjsurg.2010.07.009. PMID 21056145
- [Result] Beaver K, Latif S, Williamson S, Procter D, Sheridan J, Heath J, Susnerwala S, Luker K. An exploratory study of the follow-up care needs of patients treated for colorectal cancer. J Clin Nurs. 2010 Dec;19(23-24):3291-300. doi: 10.1111/j.1365-2702.2010.03407.x. Epub 2010 Oct 22. PMID 20964750
- [Result] Bohnenkamp SK, McDonald P, Lopez AM, Krupinski E, Blackett A. Traditional versus telenursing outpatient management of patients with cancer with new ostomies. Oncol Nurs Forum. 2004 Sep 17;31(5):1005-10. doi: 10.1188/04.ONF.1005-1010. Print 2004 Sep. PMID 15378102
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Coffey L, Mooney O, Dunne S, Sharp L, Timmons A, Desmond D, O'Sullivan E, Timon C, Gooberman-Hill R, Gallagher P. Cancer survivors' perspectives on adjustment-focused self-management interventions: a qualitative meta-synthesis. J Cancer Surviv. 2016 Dec;10(6):1012-1034. doi: 10.1007/s11764-016-0546-3. Epub 2016 May 5. PMID 27150211
- [Result] Dabirian A, Yaghmaei F, Rassouli M, Tafreshi MZ. Quality of life in ostomy patients: a qualitative study. Patient Prefer Adherence. 2010 Dec 21;5:1-5. doi: 10.2147/PPA.S14508. PMID 21311696
- [Result] Feng S, Liang Z, Zhang R, Liao W, Chen Y, Fan Y, Li H. Effects of mobile phone WeChat services improve adherence to corticosteroid nasal spray treatment for chronic rhinosinusitis after functional endoscopic sinus surgery: a 3-month follow-up study. Eur Arch Otorhinolaryngol. 2017 Mar;274(3):1477-1485. doi: 10.1007/s00405-016-4371-0. Epub 2016 Nov 7. PMID 27822702
- [Result] Fanshawe TR, Halliwell W, Lindson N, Aveyard P, Livingstone-Banks J, Hartmann-Boyce J. Tobacco cessation interventions for young people. Cochrane Database Syst Rev. 2017 Nov 17;11(11):CD003289. doi: 10.1002/14651858.CD003289.pub6. PMID 29148565
- [Result] Karabulut HK, Dinc L, Karadag A. Effects of planned group interactions on the social adaptation of individuals with an intestinal stoma: a quantitative study. J Clin Nurs. 2014 Oct;23(19-20):2800-13. doi: 10.1111/jocn.12541. Epub 2014 Jan 31. PMID 24479766
- [Result] Lee JY, Park HA, Min YH. Transtheoretical Model-based Nursing Intervention on Lifestyle Change: A Review Focused on Intervention Delivery Methods. Asian Nurs Res (Korean Soc Nurs Sci). 2015 Jun;9(2):158-67. doi: 10.1016/j.anr.2015.05.001. Epub 2015 May 13. PMID 26160246
- [Result] Lim SH, Chan SW, Lai JH, He HG. A randomized controlled trial examining the effectiveness of a STOMA psychosocial intervention programme on the outcomes of colorectal patients with a stoma: study protocol. J Adv Nurs. 2015 Jun;71(6):1310-23. doi: 10.1111/jan.12595. Epub 2014 Dec 15. PMID 25494719
- [Result] Lim SH, Chan SW, He HG. Patients' Experiences of Performing Self-care of Stomas in the Initial Postoperative Period. Cancer Nurs. 2015 May-Jun;38(3):185-93. doi: 10.1097/NCC.0000000000000158. PMID 24836957
- [Result] Lindfred H, Saalman R, Nilsson S, Sparud-Lundin C, Lepp M. Self-reported health, self-management, and the impact of living with inflammatory bowel disease during adolescence. J Pediatr Nurs. 2012 Jun;27(3):256-64. doi: 10.1016/j.pedn.2011.02.005. Epub 2011 Mar 30. PMID 22525814
- [Result] Marcus BH, Dubbert PM, Forsyth LH, McKenzie TL, Stone EJ, Dunn AL, Blair SN. Physical activity behavior change: issues in adoption and maintenance. Health Psychol. 2000 Jan;19(1S):32-41. doi: 10.1037/0278-6133.19.suppl1.32. PMID 10709946
- [Result] Raingruber B. The effectiveness of psychosocial interventions with cancer patients: an integrative review of the literature (2006-2011). ISRN Nurs. 2011;2011:638218. doi: 10.5402/2011/638218. Epub 2011 Nov 16. PMID 22191052
- [Result] Richard AA, Shea K. Delineation of self-care and associated concepts. J Nurs Scholarsh. 2011 Sep;43(3):255-64. doi: 10.1111/j.1547-5069.2011.01404.x. Epub 2011 Jul 25. PMID 21884371
- [Result] Richbourg L, Thorpe JM, Rapp CG. Difficulties experienced by the ostomate after hospital discharge. J Wound Ostomy Continence Nurs. 2007 Jan-Feb;34(1):70-9. doi: 10.1097/00152192-200701000-00011. PMID 17228210
- [Result] Rosenberg CA, Flanagan C, Brockstein B, Obel JC, Dragon LH, Merkel DE, Wade EL, Law TM, Khandekar JD, Hensing TA. Promotion of self-management for post treatment cancer survivors: evaluation of a risk-adapted visit. J Cancer Surviv. 2016 Feb;10(1):206-19. doi: 10.1007/s11764-015-0467-6. Epub 2015 Jul 16. PMID 26178325
- [Result] Spencer L, Adams TB, Malone S, Roy L, Yost E. Applying the transtheoretical model to exercise: a systematic and comprehensive review of the literature. Health Promot Pract. 2006 Oct;7(4):428-43. doi: 10.1177/1524839905278900. Epub 2006 Jul 13. PMID 16840769

DOCUMENTS (1):
  • Informed Consent Form (2011-12-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT03681821/ICF_000.pdf